CLINICAL TRIAL: NCT03889158
Title: Effect of Age and Fitness on Vascular Function and Oxidative Stress During Acute Inflammation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Elizabeth Schroeder, PhD Candidate, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1550
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-10

CONDITIONS: Aging; Inflammation
Keywords: Cardiorespiratory Fitness; Endothelial Function; Oxidative Stress
MeSH Terms: conditions — Inflammation | interventions — Typhoid-Paratyphoid Vaccines; Vi polysaccharide vaccine, typhoid; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: The vascular response to acute inflammation and oxidative stress is non-invasively assessed in individuals who are young with low fitness, older with low fitness, or older with high fitness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute Inflammation (Experimental): All participants will receive the typhoid vaccination (intramuscular injection, 0.5 mL, 1 time).
  Interventions: Biological: Typhoid Vaccine
- Ascorbic Acid (Experimental): All participants will receive ascorbic acid (Vit C) on two occasions [oral pill, 2g, 2x (baseline, during acute inflammation)].
  Interventions: Dietary Supplement: Ascorbic Acid

INTERVENTIONS:
Biological: Typhoid Vaccine — All participants will receive the typhoid vaccine.
  Other Names: Typhim Vi; Typhoid Vi Polysaccharide Vaccine
  Arms: Acute Inflammation
Dietary Supplement: Ascorbic Acid — All participants will receive ascorbic acid.
  Arms: Ascorbic Acid

SUMMARY:
This study focuses on whether high cardiorespiratory fitness in older adults has a protective effect on the vascular response to acute inflammation in comparison to low-fit older and young adults.

DETAILED DESCRIPTION:
Acute and chronic inflammation both increase cardiovascular disease risk, especially with aging, which may be due to vascular dysfunction. Aging and inflammation also lead to increased oxidative stress, which impairs vascular function. During acute inflammation, endothelial function is altered differently in younger and older adults with decreases in endothelial function in younger, but not older adults. However, cardiorespiratory fitness is cardio-protective, impacting inflammation, vascular function, and oxidative stress. During acute inflammation, moderately fit older adults exhibit similar responses to younger adults, suggesting preserved endothelial reactivity. However, whether the protective mechanism is oxidative stress has not been confirmed. Furthermore, it is undetermined whether the vascular dysfunction is further propagated down the arterial tree during acute inflammation to the microvasculature.

The aims of this research study are to determine if age and fitness moderate the vascular response to acute inflammation and to determine if antioxidant administration eliminates vascular dysfunction during acute inflammation. The results from this study will help to elucidate if fitness is a protective and preventive measure to ameliorate the detrimental cardiovascular response to acute inflammation. Thus, this study may provide health professionals with a behavioral intervention to reduce cardiovascular disease burden in the rapidly growing aging population.

ELIGIBILITY:
Inclusion Criteria:

* Males and females willing to provide informed consent
* 18-35 or 55-75 years of age
* Non-smoker
* No use of anti-inflammatory medication within last 2 weeks
* Aerobically trained (defined as performing aerobic exercise on ≥4 days/week, for ≥30 minutes, for at least the past 3 months AND a VO2max ≥75th age- and sex-specific percentile according to ACSM)
* /// OR /// Sedentary (defined as being involved in less than 30 minutes of moderately-intense physical activity per day, < 3 days/week AND a VO2max ≤ 50th age- and sex-specific percentile according to ACSM)

Exclusion Criteria:

* Body mass index >35 kg/m2
* Pregnancy, hormone replacement therapy, or peri-menopausal
* Known cardiovascular (i.e. atherosclerosis, uncontrolled hypertension, stroke, myocardial infarction, etc.), inflammatory (i.e. Crohn's disease, arthritis, etc.), or metabolic (i.e. Diabetes mellitus) disease
* Medications known to influence cardiovascular outcomes (i.e. heart rate, blood pressure, endothelial function, etc)
* Regular use of medications to reduce inflammation (NSAIDS, aspirin, steroids, etc)
* Bleeding disorders
* Illness, other vaccination, or antioxidant use within 2 weeks prior to screening
* Typhoid vaccination within previous 2 years or prior adverse reaction
* VO2max in 51st - 74th age- and sex-specific percentile according to ACSM (measured during first testing visit)
* Non-English speaking participants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Schroeder, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Integrative Physiology Laboratory, Suite 158, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the impact of COVID-19 on study recruitment, we have insufficient data to break the older adults into fit and unfit groups. These groups were thus combined into a single "Older Adults" Group.
Groups:
- Older Adults: Individuals 55-75 years of age.
- Younger Adults: Individuals 18-35 years of age
Period: Overall Study
Arm/Group | Older Adults | Younger Adults
Started | 20 | 15
Completed | 16 | 9
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Population: Analysis only completed on individuals with complete data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Adults | Younger Adults | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (5) | 24 (4) | 50 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 13 | 3 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 8 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 25
Flow-mediated dilation [Mean (Standard Deviation); unit: % change in diameter] | 3.5 (1.9) | 6.3 (3.3) | 4.5 (2.8)
Pulse wave velocity [Mean (Standard Deviation); unit: m/s] | 8.8 (2.1) | 5.6 (.4) | 7.7 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Function
Description: Flow-mediated dilation - Brachial artery vasodilator function will be noninvasively measured through assessment of brachial artery dilation using ultrasonography. The brachial artery will be imaged proximal to placement of a blood pressure cuff just below the antecubital fossa. Endothelium-dependent dilation of the brachial artery will be measured at baseline and again for 5 minutes following ischemic stimulus (inflation of a blood pressure cuff around the forearm to 250 mmHg for 5 minutes).
Time Frame: Visit 1: At [BASELINE] and 2 hours following Vit C [BASELINE+VIT C]; Visit 2 (>72 hours after Visit 1): At baseline [PRE-INFLAMMATION BASELINE]; Visit 3 (24 hours after Visit 2): At baseline [INFLAMMATION] and 2 hours following Vit C [INFLAMMATION+VIT C]
Measure: Mean (Standard Deviation); unit: % change in diameter
Arm/Group | Older Adults | Younger Adults
Number analyzed (Participants) | 16 | 9
% change in diameter
  Baseline | 2.4 (1.8) | 5.5 (3.4)
  Baseline + Vit C | 3.4 (2.7) | 5.7 (3.0)
  Pre-Inflammation Baseline | 3.4 (1.9) | 6.3 (3.3)
  Inflammation | 1.6 (1.7) | 5.8 (3.4)
  Inflammation + Vit C | 2.8 (1.9) | 6.1 (3.2)

2. Primary Outcome: Change in Oxidative Stress
Description: Oxidized low-density lipoprotein, vitamin C and total antioxidant capacity will be assessed using standard ELISAs from a venous blood draw. The analyses of the oxidized LDL and total antioxidant capacity failed. Only data on Vitamin C are presented.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Older Adults | Younger Adults
Number analyzed (Participants) | 16 | 9
ug/mL
  Baseline | 6.2 (1.2) | 4.7 (2.1)
  Baseline + Vit C | 13.3 (2.1) | 11.7 (2.9)
  Pre-Inflammation | 5.8 (1.1) | 5.4 (1.2)
  Inflammation | 6.6 (1.1) | 7.2 (4.1)
  Inflammation + Vit C | 13.4 (3.1) | 13.3 (3.0)

3. Secondary Outcome: Change in Arterial Stiffness
Description: Central pulse wave velocity - Approximately 20-sec of pressure waveforms will be collected at the brachial, common carotid, and femoral arteries using a high-fidelity strain-gauge transducer. Pulse wave velocity will be calculated from the distances between measurement points and the measured time delay between proximal (carotid) and distal (femoral) waveforms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Older Adults | Younger Adults
Number analyzed (Participants) | 16 | 9
m/s
  Baseline | 9.3 (2.0) | 5.8 (.8)
  Baseline + Vit C | 9.9 (3.0) | 5.9 (.9)
  Pre-inflammation | 8.8 (2.1) | 5.6 (.4)
  Inflammation | 8.8 (1.7) | 5.6 (.6)
  Inflammation + Vit C | 8.9 (2.1) | 5.7 (.5)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Older Adults | Younger Adults
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03889158/Prot_SAP_000.pdf